CLINICAL TRIAL: NCT03136120
Title: Study to Assess Inhaled Drug Distribution in the Distal Lung and Interstitium Using Cryobiopsy Samples From Subjects With Suspected Interstitial Lung Disease Undergoing Cryobiopsy for Clinical Reasons
Brief Title: Cryobiopsy Study to Assess Drug Distribution in Subjects With Suspected Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 205053
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Lung Diseases, Interstitial
Keywords: Ipratropium bromide; Cryobiopsy; TBCB; IPF; Transbronchial cryobiopsy; Interstitial lung disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Ipratropium; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lung biopsy samples collected from fibrotic regions of the lung using transbrochial cryobiopsy technique will be collected for this study. Endobronchial biopsy samples will also be taken. The samples will be embedded to a suitable polymer and frozen at -80 degree Celsius ready for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with suspected fibrotic ILD: Eligible subjects will receive nebulized ipratropium bromide 500 mcg for 10 minutes. The subjects will be sedated for bronchoscopic procedure as per routine practice for subjects having bronchoscopy. Cryobiopsy samples for this study will be taken after samples required for diagnosis has been taken and it is safe to do so. One to three endobronchial forceps biopsy samples will be taken from up to 5 subjects to allow comparison of proximal and distal drug distribution.
  Interventions: Drug: Ipratropium Bromide; Procedure: Flexible Bronchoscopy/Biopsy

INTERVENTIONS:
Drug: Ipratropium Bromide — Single dose of 500 mcg Ipratropium nebulizer solution will be administered to all subjects via inhalation route using nebulizer for 10 minutes. Ipratropium bromide is a clear, colorless nebulizer solution available in white plastic ampoules.
Procedure: Flexible Bronchoscopy/Biopsy — After biopsy samples required for diagnosis have been collected, additional one to two TBCB samples will be taken for this study. 3-5 endobronchial biopsy samples will be taken from up to 5 subjects to compare drug distribution in proximal and distal lung.

SUMMARY:
Interstitial lung disease (ILD) often affects distal lung, and the evaluation of drug distribution to the relevant lung compartments is essential for development of new treatment options. This single center study will utilize samples obtained by transbronchial cryobiopsy (TBCB) procedure to assess the distribution of inhaled drugs in the lungs of the subjects with fibrotic lung disease using mass spectrometry techniques. The study will have a single visit and will include approximately 20 adult subjects with suspected fibrotic ILD and requiring TBCB as part of their diagnostic assessment. This will provide TBCB samples from up to 20 subjects, up to 5 of whom may also provide endobronchial forceps biopsy samples. The study will have 3 phases including screening to check the eligibility, biopsy phase in which all subjects will receive nebulized ipratropium bromide 500 microgram (mcg) for 10 minutes immediately before undergoing bronchoscopy and follow up phase from 7 to 14 days after the procedure. Drug distribution in the lung will be assessed by analyzing biopsy samples collected using mass spectrometry and imaging techniques.

ELIGIBILITY:
Inclusion Criteria:

* 18 and above years of age inclusive, at the time of signing the informed consent.
* Subjects with suspected ILD listed for TBCB for clinical reasons following review by the ILD services at University College London Hospitals (UCLH) in whom diagnosis has remained unclear following radiological and clinical assessment.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied, may be included only if the investigator in consultation with the Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or Female.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions.

Exclusion Criteria:

* Subjects who have a known drug allergy or other contra-indication to ipratropium bromide.
* Known hypersensitivity to atropine or ipratropium bromide or any other known drug allergies that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* As a result of the medical history, physical examination or screening investigations, the physician responsible considers the subject unfit for the study.
* The subject is unable or unwilling to perform study assessments and procedures correctly.
* Subjects with a recognized co-existing respiratory disorder (other than ILD) that in the opinion of the investigator would confound the study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female subjects above 18 years of age with suspected ILD referred for TBCB for clinical reasons, as part of their diagnostic work up, will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Evaluation of the distribution of ipratropium bromide within the cryobiopsy samples | Up to Week 4
  Images and data will be generated using mass spectrometric techniques and histology to show the distribution of ipratropium bromide within the lung cryobiopsy samples taken from subjects with suspected Interstitial Lung disease.

SECONDARY OUTCOMES:
Evaluation of the distribution of ipratropium bromide within the endobronchial sample | Up to Week 4
  Images and data will be generated using mass spectrometric techniques and histology to show the distribution of ipratropium bromide within the endobronchial samples taken from subjects with suspected Interstitial Lung disease.
Distribution of ipratropium bromide in the proximal and distal lung | Up to Week 4
  1 to 3 endobronchial biopsy samples will be taken from up to 5 subjects to allow comparison of proximal and distal drug distribution.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mikolasch TA, Oballa E, Vahdati-Bolouri M, Jarvis E, Cui Y, Cahn A, Terry RL, Sahota J, Thakrar R, Marshall P, Porter JC. Mass spectrometry detection of inhaled drug in distal fibrotic lung. Respir Res. 2022 May 11;23(1):118. doi: 10.1186/s12931-022-02026-5. PMID 35546672